CLINICAL TRIAL: NCT02653638
Title: Cerebral Vasodilator Responses in Sedentary and Exercise Trained Humans
Brief Title: Blood Brain Flow and Exercise
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-0331; CVR-AAA4385 (Other: UW-Madison Study Staff); A176000 (Other: UW, Madison); EDUC/KINESIOLOGY/KINESIO (Other: UW, Madison); 4R00HL118154-03 (NIH)
Record Dates: First submitted 2015-12-22; First posted 2016-01-12 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Cerebrovascular Circulation
Keywords: Cerebral Vasodilator Function; White Matter Hyperintensity Volume; Default Mode Network Connectivity; Cognitive Function; Cardiorespiratory Fitness; Aging
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug (Experimental): Control-Hypercapnic Trials: Three stepwise CO2 elevations will be applied to the patient by adding fractional concentration of inspired CO2 (FICO2) at 2%, 4%, and 6% each time, balanced with room air. The end tidal CO2 (PetCO2) will be elevated and maintained constant for three minutes at each target level. Breath-by-breath changes in minute ventilation (VE) and PetCO2 will be measured.
  Drug-Indomethacin: Healthy volunteers, indomethacin suspension will be orally administered at 1.2 mg/kg. After drug administration, the patient will rest quietly for 90 minutes.
  Interventions: Other: Control; Drug: Indomethacin

INTERVENTIONS:
Other: Control — 1. Transcranial Doppler
  2. Blood Pressure
  3. Heart Rate
  4. Oxygen Saturation
Drug: Indomethacin — 1. Transcranial Doppler
  2. Blood Pressure
  3. Heart Rate
  4. Oxygen Saturation

SUMMARY:
Cerebral vasodilator responses to CO2 will be measured in young healthy adults, healthy sedentary older adults, and healthy exercise trained older adults. This variable will be examined before and after administering the cyclooxygenase inhibitor indomethacin, which has been shown to blunt cerebral vasodilator responses. In addition, the investigators will examine these counter-regulatory hemodynamic mechanisms to hypoperfusion caused by indomethacin.

DETAILED DESCRIPTION:
Normal aging reduces cerebral blood flow and cognitive function. Aging also appears to alter functional connectivity within the brain, which is associated with cognitive functioning. Observational studies suggest that regular physical activity is associated with higher cerebral blood flow and improved cognitive function. However, the mechanistic links among regular physical activity and cerebral blood flow with advancing age are unknown. In this context, it is unclear if aging or exercise training status alters the neurovascular coupling of blood flow in the brain. Thus, the overall goal of this study is to examine the age-related changes in cerebral vasodilatory capacity, an important homeostatic mechanism and marker for effective regulation of cerebral perfusion, in order to determine how it is mechanistically linked to cognition. Additionally, the investigators will explore the potential beneficial effect of physical activity on the relationships between cerebral vasodilation and cognition in humans.

The research aims are:

1. To determine if cerebral vasodilator responses are affected by age and exercise training status in healthy adults.
2. To compare the effect of cyclooxygenase inhibition on cerebral vasodilator responses in healthy adults.
3. To determine the neurovascular counter-regulatory response to cyclooxygenase inhibition in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Young subjects between 18-35 years old
* Older subjects between 55-75 years old
* Nonsmokers
* Physically active (exercise more than 3 times per week for at least 30 minutes)
* Sedentary (no formal exercise over 1 hour per week).

Exclusion Criteria:

* Outside of the specified age range
* Present with history or evidence of hepatic, renal, or hematological disease; peripheral vascular disease; stroke/neurovascular disease; diabetes; hypertension
* Take medications that indicate hepatic, renal, hematological disease; cardiovascular disease, including hypertension; stroke/neurovascular disease; and diabetes
* Body mass index >34 kg/m2
* Take physician-prescribed medications that may interact with indomethacin: 1) cardiovascular drugs (e.g. angiotensin-converting-enzyme inhibitor (ACE inhibitors), angiotensin II receptor blockers (ARB's), Diuretics); 2) drugs that would increase bleeding risk (e.g. warfarin, heparin, clopidogrel, rivaroxaban, other NSAIDs); or 3) drugs associated with increased renal toxicity (e.g. cyclosporin, tacrolimus)
* Vulnerable populations (i.e. pregnant women, prisoners, individuals lacking capacity to consent, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Cerebral Vasodilator Responses | Measurement at baseline
  Utilize a Transcranial Doppler to measure blood flow velocity in response to inhaled carbon dioxide.

SECONDARY OUTCOMES:
Cerebral Vasodilator Responses | Measurement beginning 60 minutes post drug and measured through 180 minutes
  Utilize a Transcranial Doppler to measure blood flow velocity in response to inhaled carbon dioxide.
Blood Pressure | Measurement at baseline and beginning 60 minutes post drug and measured through 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jill N Barnes, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Gymnasium-Natatorium, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews-Hanna JR, Snyder AZ, Vincent JL, Lustig C, Head D, Raichle ME, Buckner RL. Disruption of large-scale brain systems in advanced aging. Neuron. 2007 Dec 6;56(5):924-35. doi: 10.1016/j.neuron.2007.10.038. PMID 18054866
- [Background] Damoiseaux JS, Beckmann CF, Arigita EJ, Barkhof F, Scheltens P, Stam CJ, Smith SM, Rombouts SA. Reduced resting-state brain activity in the "default network" in normal aging. Cereb Cortex. 2008 Aug;18(8):1856-64. doi: 10.1093/cercor/bhm207. Epub 2007 Dec 5. PMID 18063564
- [Background] Ainslie PN, Cotter JD, George KP, Lucas S, Murrell C, Shave R, Thomas KN, Williams MJ, Atkinson G. Elevation in cerebral blood flow velocity with aerobic fitness throughout healthy human ageing. J Physiol. 2008 Aug 15;586(16):4005-10. doi: 10.1113/jphysiol.2008.158279. Epub 2008 Jul 17. PMID 18635643
- [Background] Erickson KI, Voss MW, Prakash RS, Basak C, Szabo A, Chaddock L, Kim JS, Heo S, Alves H, White SM, Wojcicki TR, Mailey E, Vieira VJ, Martin SA, Pence BD, Woods JA, McAuley E, Kramer AF. Exercise training increases size of hippocampus and improves memory. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3017-22. doi: 10.1073/pnas.1015950108. Epub 2011 Jan 31. PMID 21282661
- [Background] Bakker SL, de Leeuw FE, den Heijer T, Koudstaal PJ, Hofman A, Breteler MM. Cerebral haemodynamics in the elderly: the rotterdam study. Neuroepidemiology. 2004 Jul-Aug;23(4):178-84. doi: 10.1159/000078503. PMID 15272220
- [Background] Selim M, Jones R, Novak P, Zhao P, Novak V. The effects of body mass index on cerebral blood flow velocity. Clin Auton Res. 2008 Dec;18(6):331-8. doi: 10.1007/s10286-008-0490-z. Epub 2008 Aug 22. PMID 18726054
- [Background] Dandona P, James IM, Newbury PA, Woollard ML, Beckett AG. Cerebral blood flow in diabetes mellitus: evidence of abnormal cerebrovascular reactivity. Br Med J. 1978 Jul 29;2(6133):325-6. doi: 10.1136/bmj.2.6133.325. PMID 687900
- [Background] Barnes JN, Schmidt JE, Nicholson WT, Joyner MJ. Cyclooxygenase inhibition abolishes age-related differences in cerebral vasodilator responses to hypercapnia. J Appl Physiol (1985). 2012 Jun;112(11):1884-90. doi: 10.1152/japplphysiol.01270.2011. Epub 2012 Mar 22. PMID 22442028
- [Background] Lipsitz LA, Mukai S, Hamner J, Gagnon M, Babikian V. Dynamic regulation of middle cerebral artery blood flow velocity in aging and hypertension. Stroke. 2000 Aug;31(8):1897-903. doi: 10.1161/01.str.31.8.1897. PMID 10926954
- [Background] Kearney-Schwartz A, Rossignol P, Bracard S, Felblinger J, Fay R, Boivin JM, Lecompte T, Lacolley P, Benetos A, Zannad F. Vascular structure and function is correlated to cognitive performance and white matter hyperintensities in older hypertensive patients with subjective memory complaints. Stroke. 2009 Apr;40(4):1229-36. doi: 10.1161/STROKEAHA.108.532853. Epub 2009 Feb 26. PMID 19246701
- [Background] Smith EE, Greenberg SM. Beta-amyloid, blood vessels, and brain function. Stroke. 2009 Jul;40(7):2601-6. doi: 10.1161/STROKEAHA.108.536839. Epub 2009 May 14. PMID 19443808
- [Background] Girouard H, Iadecola C. Neurovascular coupling in the normal brain and in hypertension, stroke, and Alzheimer disease. J Appl Physiol (1985). 2006 Jan;100(1):328-35. doi: 10.1152/japplphysiol.00966.2005. PMID 16357086
- [Background] Celermajer DS, Sorensen KE, Bull C, Robinson J, Deanfield JE. Endothelium-dependent dilation in the systemic arteries of asymptomatic subjects relates to coronary risk factors and their interaction. J Am Coll Cardiol. 1994 Nov 15;24(6):1468-74. doi: 10.1016/0735-1097(94)90141-4. PMID 7930277
- [Background] Panza JA, Quyyumi AA, Brush JE Jr, Epstein SE. Abnormal endothelium-dependent vascular relaxation in patients with essential hypertension. N Engl J Med. 1990 Jul 5;323(1):22-7. doi: 10.1056/NEJM199007053230105. PMID 2355955
- [Background] Kugiyama K, Kerns SA, Morrisett JD, Roberts R, Henry PD. Impairment of endothelium-dependent arterial relaxation by lysolecithin in modified low-density lipoproteins. Nature. 1990 Mar 8;344(6262):160-2. doi: 10.1038/344160a0. PMID 2106627
- [Background] Luscher TF, Diederich D, Siebenmann R, Lehmann K, Stulz P, von Segesser L, Yang ZH, Turina M, Gradel E, Weber E, et al. Difference between endothelium-dependent relaxation in arterial and in venous coronary bypass grafts. N Engl J Med. 1988 Aug 25;319(8):462-7. doi: 10.1056/NEJM198808253190802. PMID 3136329
- [Background] Taddei S, Virdis A, Ghiadoni L, Versari D, Salvetti A. Which endothelium-derived factors are really important in humans? Biol Chem. 2006 Feb;387(2):151-7. doi: 10.1515/BC.2006.020. PMID 16497146
- [Background] Taddei S, Virdis A, Mattei P, Ghiadoni L, Gennari A, Fasolo CB, Sudano I, Salvetti A. Aging and endothelial function in normotensive subjects and patients with essential hypertension. Circulation. 1995 Apr 1;91(7):1981-7. doi: 10.1161/01.cir.91.7.1981. PMID 7895356
- [Background] Mitchell GF, van Buchem MA, Sigurdsson S, Gotal JD, Jonsdottir MK, Kjartansson O, Garcia M, Aspelund T, Harris TB, Gudnason V, Launer LJ. Arterial stiffness, pressure and flow pulsatility and brain structure and function: the Age, Gene/Environment Susceptibility--Reykjavik study. Brain. 2011 Nov;134(Pt 11):3398-407. doi: 10.1093/brain/awr253. PMID 22075523
- [Background] Ide K, Eliasziw M, Poulin MJ. Relationship between middle cerebral artery blood velocity and end-tidal PCO2 in the hypocapnic-hypercapnic range in humans. J Appl Physiol (1985). 2003 Jul;95(1):129-37. doi: 10.1152/japplphysiol.01186.2002. PMID 19278048
- [Background] Ivancev V, Bakovic D, Obad A, Breskovic T, Palada I, Joyner MJ, Dujic Z. Effects of indomethacin on cerebrovascular response to hypercapnea and hypocapnea in breath-hold diving and obstructive sleep apnea. Respir Physiol Neurobiol. 2009 May 15;166(3):152-8. doi: 10.1016/j.resp.2009.03.001. Epub 2009 Mar 18. PMID 19442931
- [Background] Xie A, Skatrud JB, Morgan B, Chenuel B, Khayat R, Reichmuth K, Lin J, Dempsey JA. Influence of cerebrovascular function on the hypercapnic ventilatory response in healthy humans. J Physiol. 2006 Nov 15;577(Pt 1):319-29. doi: 10.1113/jphysiol.2006.110627. Epub 2006 Aug 24. PMID 16931556
- [Background] DeSouza CA, Shapiro LF, Clevenger CM, Dinenno FA, Monahan KD, Tanaka H, Seals DR. Regular aerobic exercise prevents and restores age-related declines in endothelium-dependent vasodilation in healthy men. Circulation. 2000 Sep 19;102(12):1351-7. doi: 10.1161/01.cir.102.12.1351. PMID 10993851
- [Background] Kelley RE, Chang JY, Scheinman NJ, Levin BE, Duncan RC, Lee SC. Transcranial Doppler assessment of cerebral flow velocity during cognitive tasks. Stroke. 1992 Jan;23(1):9-14. doi: 10.1161/01.str.23.1.9. PMID 1731426
- [Background] Droste DW, Harders AG, Rastogi E. A transcranial Doppler study of blood flow velocity in the middle cerebral arteries performed at rest and during mental activities. Stroke. 1989 Aug;20(8):1005-11. doi: 10.1161/01.str.20.8.1005. PMID 2667197
- [Background] Geda YE, Roberts RO, Knopman DS, Christianson TJ, Pankratz VS, Ivnik RJ, Boeve BF, Tangalos EG, Petersen RC, Rocca WA. Physical exercise, aging, and mild cognitive impairment: a population-based study. Arch Neurol. 2010 Jan;67(1):80-6. doi: 10.1001/archneurol.2009.297. PMID 20065133
- [Background] Baker LD, Frank LL, Foster-Schubert K, Green PS, Wilkinson CW, McTiernan A, Cholerton BA, Plymate SR, Fishel MA, Watson GS, Duncan GE, Mehta PD, Craft S. Aerobic exercise improves cognition for older adults with glucose intolerance, a risk factor for Alzheimer's disease. J Alzheimers Dis. 2010;22(2):569-79. doi: 10.3233/JAD-2010-100768. PMID 20847403
- [Background] Lautenschlager NT, Cox KL, Flicker L, Foster JK, van Bockxmeer FM, Xiao J, Greenop KR, Almeida OP. Effect of physical activity on cognitive function in older adults at risk for Alzheimer disease: a randomized trial. JAMA. 2008 Sep 3;300(9):1027-37. doi: 10.1001/jama.300.9.1027. PMID 18768414
- [Background] Galetta F, Franzoni F, Plantinga Y, Ghiadoni L, Rossi M, Prattichizzo F, Carpi A, Taddei S, Santoro G. Ambulatory blood pressure monitoring and endothelium-dependent vasodilation in the elderly athletes. Biomed Pharmacother. 2006 Sep;60(8):443-7. doi: 10.1016/j.biopha.2006.07.013. Epub 2006 Aug 2. PMID 16904861
- [Background] Franzoni F, Ghiadoni L, Galetta F, Plantinga Y, Lubrano V, Huang Y, Salvetti G, Regoli F, Taddei S, Santoro G, Salvetti A. Physical activity, plasma antioxidant capacity, and endothelium-dependent vasodilation in young and older men. Am J Hypertens. 2005 Apr;18(4 Pt 1):510-6. doi: 10.1016/j.amjhyper.2004.11.006. PMID 15831361
- [Background] Green DJ, O'Driscoll G, Joyner MJ, Cable NT. Exercise and cardiovascular risk reduction: time to update the rationale for exercise? J Appl Physiol (1985). 2008 Aug;105(2):766-8. doi: 10.1152/japplphysiol.01028.2007. Epub 2008 Jan 3. No abstract available. PMID 18174390
- [Background] Seifert T, Brassard P, Wissenberg M, Rasmussen P, Nordby P, Stallknecht B, Adser H, Jakobsen AH, Pilegaard H, Nielsen HB, Secher NH. Endurance training enhances BDNF release from the human brain. Am J Physiol Regul Integr Comp Physiol. 2010 Feb;298(2):R372-7. doi: 10.1152/ajpregu.00525.2009. Epub 2009 Nov 18. PMID 19923361
- [Background] Serrador JM, Picot PA, Rutt BK, Shoemaker JK, Bondar RL. MRI measures of middle cerebral artery diameter in conscious humans during simulated orthostasis. Stroke. 2000 Jul;31(7):1672-8. doi: 10.1161/01.str.31.7.1672. PMID 10884472
- [Background] Raz L, Jayachandran M, Tosakulwong N, Lesnick TG, Wille SM, Murphy MC, Senjem ML, Gunter JL, Vemuri P, Jack CR Jr, Miller VM, Kantarci K. Thrombogenic microvesicles and white matter hyperintensities in postmenopausal women. Neurology. 2013 Mar 5;80(10):911-8. doi: 10.1212/WNL.0b013e3182840c9f. Epub 2013 Feb 13. PMID 23408873
- [Background] MacLeod CM. Half a century of research on the Stroop effect: an integrative review. Psychol Bull. 1991 Mar;109(2):163-203. doi: 10.1037/0033-2909.109.2.163. No abstract available. PMID 2034749
- [Background] Lucas SJ, Ainslie PN, Murrell CJ, Thomas KN, Franz EA, Cotter JD. Effect of age on exercise-induced alterations in cognitive executive function: relationship to cerebral perfusion. Exp Gerontol. 2012 Aug;47(8):541-51. doi: 10.1016/j.exger.2011.12.002. Epub 2012 Jan 2. PMID 22230488
- [Background] Owen AM, Downes JJ, Sahakian BJ, Polkey CE, Robbins TW. Planning and spatial working memory following frontal lobe lesions in man. Neuropsychologia. 1990;28(10):1021-34. doi: 10.1016/0028-3932(90)90137-d. PMID 2267054
- [Background] Frauenfelder BA, Schuepbach D, Baumgartner RW, Hell D. Specific alterations of cerebral hemodynamics during a planning task: a transcranial Doppler sonography study. Neuroimage. 2004 Jul;22(3):1223-30. doi: 10.1016/j.neuroimage.2004.03.008. PMID 15219594
- [Background] Schuepbach D, Boeker H, Duschek S, Hell D. Rapid cerebral hemodynamic modulation during mental planning and movement execution: evidence of time-locked relationship with complex behavior. Clin Neurophysiol. 2007 Oct;118(10):2254-62. doi: 10.1016/j.clinph.2007.07.013. Epub 2007 Sep 4. PMID 17766175
- [Background] Jensen K, Kjaergaard S, Malte E, Bunemann L, Therkelsen K, Knudsen F. Effect of graduated intravenous and standard rectal doses of indomethacin on cerebral blood flow in healthy volunteers. J Neurosurg Anesthesiol. 1996 Apr;8(2):111-6. doi: 10.1097/00008506-199604000-00002. PMID 8829556
- [Background] Carlsson I, Wennmalm A. Effect of different prostaglandin synthesis inhibitors on post-occlusive blood flow in human forearm. Prostaglandins. 1983 Aug;26(2):241-52. doi: 10.1016/0090-6980(83)90092-8. PMID 6417728